CLINICAL TRIAL: NCT02053610
Title: An Open-label, Multi-center, Three Arm Randomized Study to Investigate the Safety and Efficacy on Progression-free Survival of RO5072759 + Chlorambucil (GClb) Compared to Rituximab + Chlorambucil (RClb) or Chlorambucil (Clb) Alone in Previously Untreated CLL Patients With Comorbidities.
Brief Title: CLL11: A Study of Obinutuzumab (RO5072759 [GA101]) With Chlorambucil in Patients With Previously Untreated Chronic Lymphocytic Leukemia (Stage 2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: German CLL Study Group (Other); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO21004 (Stage 2); 2009-012476-28; CLL1
Record Dates: First submitted 2013-11-25; First posted 2014-02-03 (Estimated); Results first posted 2014-10-10 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-08

CONDITIONS: Lymphocytic Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — obinutuzumab; Rituximab; Chlorambucil

ARMS (3):
- obinutuzumab + chlorambucil (GClb) (Experimental): Participants received 1000 mg obinutuzumab intravenous (IV) infusion, on Days 1 [first infusion split 100 mg on Day 1 and 900 mg on Day 2 as per protocol amendment], 8 and 15 in Cycle 1 and Day 1 in Cycles 2-6 (28-day cycles) plus chlorambucil 0.5 mg/kg orally on Day 1 and 15 of each 28-day cycle (6 Cycles).
  Interventions: Drug: obinutuzumab; Drug: chlorambucil
- rituximab + chlorambucil (RClb) (Active Comparator): Participants received 375 mg/m^2 rituximab IV infusion on Day 1 of Cycle 1 then 500 mg/m^2 IV infusions on Day 1 of Cycles 2-6 (28-day cycles) plus chlorambucil 0.5 mg/kg orally on Day 1 and 15 of each 28-day cycle (6 cycles).
  Interventions: Drug: rituximab; Drug: chlorambucil
- Chlorambucil (Clb) (Active Comparator): Participants received chlorambucil 0.5 mg/kg orally on Day 1 and 15 of each 28-day cycle (6 Cycles). Participants with Progressive Disease or within 6 months of follow-up were allowed to cross over to receive obinutuzumab + chlorambucil.
  Interventions: Drug: chlorambucil

INTERVENTIONS:
Drug: obinutuzumab — 1000 mg obinutuzumab intravenous (IV) infusion, on Days 1 [first infusion split 100 mg on Day 1 and 900 mg on Day 2 as per protocol amendment], 8 and 15 in Cycle 1 and Day 1 in Cycles 2-6 (28-day cycles).
  Other Names: RO5072759; GA101; GAZYVA®; Gazyvaro
  Arms: obinutuzumab + chlorambucil (GClb)
Drug: rituximab — 375 mg/m^2 rituximab intravenous (IV) infusion on Day 1 of Cycle 1 (Cycle duration is 28 days) then 500 mg/m^2 IV infusions on Day 1 of Cycles 2-6.
  Other Names: Rituxan®; MabThera®
  Arms: rituximab + chlorambucil (RClb)
Drug: chlorambucil — Chlorambucil 0.5 mg/kg orally on Day 1 and 15 of each 28-day cycle

SUMMARY:
This open-label, randomized, 3-arm study will evaluate the efficacy and safety of (obinutuzumab) RO5072759 in combination with chlorambucil as compared to rituximab plus chlorambucil or chlorambucil alone in patients with previously untreated chronic lymphocytic leukemia (CLL). Patients will be randomized 2:2:1 to receive a maximum of six 28-day cycles of either RO5072759 (1000 mg intravenous (iv) infusion, on days 1, 8 and 15 of cycle 1 and day 1 of cycles 2-6) plus chlorambucil (0.5 mg/kg orally, days 1 and 15 of cycles 1-6), or rituximab (iv infusion day 1, 375 mg/m^2 cycle 1, 500 mg/m^2 cycles 2-6) plus chlorambucil, or chlorambucil alone. Anticipated time on study treatment is >6 months and follow-up for disease-progression and safety will be at least 5 years. In the US, this trial is sponsored/managed by Genentech.

DETAILED DESCRIPTION:
Protocol BO21004 is divided into 3 separate Unique Protocol IDs for reporting results on clinicaltrials.gov because there are 3 separate primary analyses conducted at different time-points.

* BO21004 (Stage 1a) [NCT01010061] includes the analysis of 2 of the 3 arms obinutuzumab plus chlorambucil (Glb) compared to chlorambucil (Clb) reported separately.
* BO21004 (Stage 1b) [NCT01998880] includes the analysis of 2 of the 3 arms rituximab plus chlorambucil (RClb) compared to chlorambucil (Clb) reported separately.
* BO21004 (Stage 2) includes the analysis of 2 of the 3 arms obinutuzumab plus chlorambucil (Glb) compared to rituximab plus chlorambucil (RClb) reported here.

ELIGIBILITY:
Inclusion Criteria:

* Adults >/=18 years
* Documented Cluster of Differentiation Antigen 20 (CD20) + B-Cell Chronic Lymphocytic Lymphoma (B-CLL)
* Previously untreated Chronic Lymphocytic Leukemia (CLL) requiring treatment according to the National Cancer Institute (NCI) criteria
* Total Cumulative Illness Rating Scale (CIRS) > 6 and/or creatinine clearance < 70 ml/min.

Exclusion Criteria:

* Prior CLL therapy
* Transformation of CLL to aggressive Non-Hodgkin's Lymphoma (NHL) (Richter's transformation)
* History of other malignancy unless the malignancy has been in remission without treatment for >/=2 years prior to enrolment, and except for carcinoma in situ of the cervix, basal or squamous cell skin cancer, surgically treated low-grade prostate cancer, or ductal carcinoma in situ (DCIS) of the breast treated with lumpectomy alone
* Positive hepatitis serology (HBV, HCV) or positive HIV or Human T-Cell Leukemia Virus (HTLV) testing
* Patients with active infection requiring systemic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 787 (Actual)
Dates: Start 2009-12-31 (Actual); Primary Completion 2013-08-31 (Actual); Study Completion 2017-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (214):
- United States (5):
  - San Diego, California
  - Chicago, Illinois
  - Baltimore, Maryland
  - Green Bay, Wisconsin
  - Waukesha, Wisconsin
- Argentina (2):
  - Buenos Aires
  - Rosario
- Australia (12):
  - Adelaide, New South Wales
  - Gosford, New South Wales
  - Kogarah, New South Wales
  - Liverpool, New South Wales
  - St Leonards, New South Wales
  - Sydney, New South Wales
  - Greenslopes, Queensland
  - Southport, Queensland
  - Woolloongabba, Queensland
  - Kurralta Park, South Australia
  - Frankston, Victoria
  - Melbourne, Victoria
- Austria (3):
  - Graz
  - Innsbruck
  - Vienna
- Brazil (5):
  - Goiânia, Goiás
  - Belo Horizonte, Minas Gerais
  - Porto Alegre, Rio Grande do Sul
  - Santo André, São Paulo
  - São Paulo, São Paulo
- Bulgaria (5):
  - Pleven
  - Plovdiv
  - Sofia
  - Varna
  - Vratsa
- Canada (8):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - Barrie, Ontario
  - Ottawa, Ontario
  - Montreal, Quebec
  - Rimouski, Quebec
- Zagreb, Croatia
- Czechia (3):
  - Brno
  - Hradec Králové
  - Prague
- Denmark (5):
  - Aalborg
  - Aarhus
  - Copenhagen
  - Odense
  - Vejle
- Cairo, Egypt
- Estonia (2):
  - Tallinn
  - Tartu
- France (21):
  - Angers
  - Bobigny
  - Caen
  - Clermont-Ferrand
  - Créteil
  - Le Mans
  - Lille
  - Lyon
  - Marseille
  - Montpellier
  - Nantes
  - Paris
  - Pessac
  - Pierre-Bénite
  - Poitiers
  - Reims
  - Rennes
  - Rouen
  - Toulouse
  - Tours
  - Vandœuvre-lès-Nancy
- Germany (67):
  - Ahaus
  - Amberg
  - Ansbach
  - Bamberg
  - Berlin
  - Bonn
  - Bremen
  - Cologne
  - Delitzsch
  - Detmold
  - Dresden
  - Duisburg
  - Erlangen
  - Eschweiler
  - Essen
  - Esslingen am Neckar
  - Frankfurt
  - Frankfurt (Oder)
  - Frankfurt am Main
  - Frechen
  - Freiburg im Breisgau
  - Giessen
  - Göttingen
  - Greifswald
  - Hamburg
  - Hamm
  - Hanover
  - Heidelberg
  - Homburg/Saar
  - Kaiserslautern
  - Karlsruhe
  - Kempten
  - Kiel
  - Koblenz
  - Kronach
  - Landshut
  - Lebach
  - Leer
  - Lemgo
  - Loerrach
  - Lüdenscheid
  - Magedburg
  - Mainz
  - Mannheim
  - Mutlangen
  - München
  - Neunkirchen/Saar
  - Nuremberg
  - Oldenburg
  - Porta Westfalica
  - Ravensburg
  - Recklinghausen
  - Regensburg
  - Rostock
  - Rüsselsheim am Main
  - Saarbrücken
  - Sindelfingen
  - Stuttgart
  - Trier
  - Tübingen
  - Ulm
  - Villingen-Schwenningen
  - Weilheim
  - Wendlingen
  - Witten
  - Worms
  - Würzburg
- Hong Kong, Hong Kong
- Italy (11):
  - Cosenza, Calabria
  - Ferrara, Emilia-Romagna
  - Modena, Emilia-Romagna
  - Rome, Lazio
  - Genoa, Liguria
  - Milan, Lombardy
  - Orbassano, Piedmont
  - Turin, Piedmont
  - Cagliari, Sardinia
  - Messina, Sicily
  - Terni, Umbria
- Mexico (5):
  - Aguascalientes
  - Culiacán
  - Hermosillo
  - Monterrey
  - San Luis Potosí City
- Netherlands (4):
  - Delftzijl
  - Enschede
  - Leeuwarden
  - Nieuwegein
- New Zealand (2):
  - Auckland
  - Christchurch
- Romania (2):
  - Bucharest
  - Târgu Mureş
- Russia (6):
  - Kazan'
  - Nizhny Novgorod
  - Penza
  - Perm
  - Rostov-on-Don
  - Ufa
- Bratislava, Slovakia
- Spain (22):
  - Manresa, Barcelona
  - Sabadell, Barcelona
  - Jerez de la Frontera, Cadiz
  - Santander, Cantabria
  - Donostia / San Sebastian, Guipuzcoa
  - A Coruña, LA Coruña
  - Santiago de Compostela, LA Coruña
  - Pamplona, Navarre
  - Oviedo, Principality of Asturias
  - San Cristóbal de La Laguna, Tenerife
  - Gandia, Valencia
  - Barcelona
  - Jaén
  - Las Palmas
  - Madrid
  - Málaga
  - Murcia
  - Salamanca
  - Seville
  - Toledo
  - Valencia
  - Zaragoza
- Switzerland (7):
  - Aarau
  - Basel
  - Bern
  - Chur
  - Lucerne
  - Sankt Gallen
  - Zurich
- Thailand (2):
  - Bangkok
  - Khon Kaen
- United Kingdom (11):
  - Bournemouth
  - Cambridge
  - Canterbury
  - Cardiff
  - Cottingham
  - Edinburgh
  - Glasgow
  - Leicester
  - London
  - Nottingham
  - Sutton

REFERENCES:
- [Derived] Dimier N, Delmar P, Ward C, Morariu-Zamfir R, Fingerle-Rowson G, Bahlo J, Fischer K, Eichhorst B, Goede V, van Dongen JJM, Ritgen M, Bottcher S, Langerak AW, Kneba M, Hallek M. A model for predicting effect of treatment on progression-free survival using MRD as a surrogate end point in CLL. Blood. 2018 Mar 1;131(9):955-962. doi: 10.1182/blood-2017-06-792333. Epub 2017 Dec 18. PMID 29255066

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 787 patients were enrolled in the study. Following a 6 patient safety run-in prior to randomization, 781 patients were randomized.
Pre-assignment Details: 589 patients were randomized to 1 of 3 treatment groups in 2:2:1 ratio: GClb (n=238), RClb (n=233) or Clb (n=118) in Stage 1 and an additional 192 randomized to GClb or RClb in Stage 2. Stage 1 was divided for analysis into: Stage 1a [NCT01010061] and Stage 1b [NCT01998880]. 663 participants were included in the Stage 2 Analysis reported here.
Period: Overall Study
Arm/Group | Rituximab + Chlorambucil (RClb) | Obinutuzumab + Chlorambucil (GClb)
Started | 330 | 333
Received Study Drug | 326 | 331
Completed | 288 (Completed=Completed Treatment) | 266 (Completed=Completed Treatment)
Not Completed | 42 | 67
Not completed — Adverse Event/Intercurrent Illness | 25 | 43
Not completed — Withdrew Consent | 2 | 9
Not completed — Death | 5 | 5
Not completed — Administrative/Other | 1 | 1
Not completed — Disease Progression | 2 | 3
Not completed — Refused treatment/Did not cooperate | 1 | 3
Not completed — Did not Receive Treatment | 4 | 2
Not completed — Insufficient Therapeutic Response | 1 | 1
Not completed — Violation of Selection Criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab + Chlorambucil (RClb) | Obinutuzumab + Chlorambucil (GClb) | Total
Number analyzed (Participants) | 330 | 333 | 663
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (8.82) | 71.9 (8.68) | 71.7 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 130 | 256
  Male | 204 | 203 | 407

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from randomization to the first occurrence of progression, relapse, or death from any cause as assessed by the investigator. Progressive disease required at least one of the following: ≥50% increase in the absolute number of lymphocytes, appearance of new palpable lymph nodes (>15 mm in longest diameter) or any new extra nodal lesion, ≥50% increase in the longest diameter of any previous site of clinically significant lymphadenopathy, ≥50% increase in the enlargement of the liver and/or spleen, Transformation to a more aggressive histology or After treatment, the progression of any cytopenia (a decrease of hemoglobin levels >20 g/L or <10 g/dL or a decrease of platelet counts >50% or <100 x 10^9/L or by a decrease of neutrophil counts >50% or <1.0 x 10^9/L).
Time Frame: Randomization to clinical cutoff (median observation 59.4 months)
Population: Intent--to-treat population (ITT) included all randomized participants. Data for patients without disease progression or death was censored at the time of the last response assessment, or, if no response assessments were performed after the baseline visit, at the time of randomization plus one day.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab + Chlorambucil (RClb) | Obinutuzumab + Chlorambucil (GClb)
Number analyzed (Participants) | 330 | 333
months | 15.7 [14.3 to 17.2] | 28.9 [26.1 to 32.7]
Statistical Analysis 1: Comparison: Rituximab + Chlorambucil (RClb) vs Obinutuzumab + Chlorambucil (GClb); Test type: Superiority or Other; p < 0.0001, Log Rank, Stratified; Stratified by Binet stage at Baseline; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.41 to 0.58]

2. Primary Outcome: Percentage of Participants With Progression Free Survival Events
Description: Percentage of Participants with Progression Free Survival Events: progression, relapse, or death.
Time Frame: Randomization to clinical cutoff (median observation 59.4 months)
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Chlorambucil (RClb) | Obinutuzumab + Chlorambucil (GClb)
Number analyzed (Participants) | 330 | 333
percentage of participants | 88.5 | 73.3

3. Secondary Outcome: Progression Free Survival Based on Independent Review Committee (IRC) Data
Description: PFS was defined as the time from randomization to the first occurrence of progression, relapse, or death from any cause as assessed by Independent Review Committee. Progressive disease required at least one of the following: ≥50% increase in the absolute number of lymphocytes, appearance of new palpable lymph nodes (>15 mm in longest diameter) or any new extra nodal lesion, ≥50% increase in the longest diameter of any previous site of clinically significant lymphadenopathy, ≥50% increase in the enlargement of the liver and/or spleen, Transformation to a more aggressive histology or After treatment, the progression of any cytopenia (a decrease of hemoglobin levels >20 g/L or <10 g/dL or a decrease of platelet counts >50% or <100 x 10^9/L or by a decrease of neutrophil counts >50% or <1.0 x 10^9/L).
Time Frame: Randomization to clinical cutoff of 09 May 2013 (median observation 18.7 months)
Population: Intent-to-treat population (ITT) included all randomized participants. Data for patients without disease progression or death was censored at the time of the last response assessment, or, if no response assessments were performed after the baseline visit, at the time of randomization plus one day.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab + Chlorambucil (RClb) | Obinutuzumab + Chlorambucil (GClb)
Number analyzed (Participants) | 330 | 333
months | 14.9 [14.2 to 17.2] | 26.7 [23.2 to 31.1]
Statistical Analysis 1: Comparison: Rituximab + Chlorambucil (RClb) vs Obinutuzumab + Chlorambucil (GClb); Test type: Superiority or Other; p < 0.0001, Log Rank, Stratified; Stratified by Binet stage at Baseline; Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.33 to 0.54] — Stratified by Binet stage at Baseline

4. Secondary Outcome: Percentage of Participants With Progression Free Survival Events Based on Independent Review Committee (IRC) Data
Description: Percentage of Participants with Progression Free Survival Events: progression, relapse, or death from any cause as assessed by an Independent Review Committee.
Time Frame: Randomization to clinical cutoff of 09 May 2013 (median observation 18.7 months)
Population: ITT participants included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Chlorambucil (RClb) | Obinutuzumab + Chlorambucil (GClb)
Number analyzed (Participants) | 330 | 333
percentage of participants | 55.5 | 30.9

5. Secondary Outcome: Percentage of Participants With End of Treatment Response (EOTR)
Description: EOTR was the first response assessment 56 days from the last dose according to the International Workshop on Chronic Lymphocytic Leukaemia (IWCLL) guidelines. Complete Response (CR) required: Peripheral blood lymphocytes below 4 x 10^9/L, Absence of significant lymphadenopathy, No hepatomegaly, No splenomegaly, Absence of disease, Blood counts above the following values (Neutrophils >1.5 x 10^9/L, Platelets >100 x 10^9/L, Hemoglobin >11g/dL) and Bone marrow at least normocellular for age. CRi was CR with incomplete bone marrow recovery. Partial Response (PR) required the following for at least 2 months from end of treatment: ≥50% decrease in peripheral blood lymphocyte count from the pre-treatment value AND Either a ≥ 50% reduction in lymphadenopathy OR ≥50% reduction of liver enlargement OR ≥50% reduction of spleen enlargement PLUS at least one of the following: Neutrophils >1.5 x 10^9/ or ≥50% increase, Platelets >100 x 10^9/L or ≥50% increase, Hemoglobin 11 g/dL or ≥50% increase.
Time Frame: Randomization to clinical cutoff (median observation 59.4 months)
Population: Participants from the ITT population, all randomized participants, with data available for analysis. Participants who had not reached the 3-month follow-up visit at the time of the clinical cut-off were excluded from analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab + Chlorambucil (RClb) | Obinutuzumab + Chlorambucil (GClb)
Number analyzed (Participants) | 330 | 333
percentage of participants
  Complete Response (CR) | 4.8 [2.8 to 7.8] | 15.6 [11.9 to 20]
  Complete Response incomplete (CRi) | 1.5 [0.5 to 3.5] | 3.6 [1.9 to 6.2]
  Partial Response (PR) | 53.9 [48.4 to 59.4] | 52.0 [46.4 to 57.4]
  Nodular Partial Response (nPR) | 5.2 [3.0 to 8.1] | 7.5 [4.9 to 10.9]
  Stable Disease | 15.2 [11.5 to 19.5] | 4.5 [2.5 to 7.3]
  Progressive Disease | 11.2 [8.0 to 15.1] | 4.5 [2.5 to 7.3]
  No Response Assessment | 8.2 [NA to NA] — 95% CI not estimated for No Response Assessment category. | 12.3 [NA to NA] — 95% CI not estimated for No Response Assessment category.
Statistical Analysis 1: Comparison: Rituximab + Chlorambucil (RClb) vs Obinutuzumab + Chlorambucil (GClb); Includes participants with EOTR: CR, CRi, PR or nPR; Test type: Superiority or Other; p = 0.0001, Chi-squared; Difference in Response Rates = 13.22, 95% CI 2-sided [6.3 to 20.1]

6. Secondary Outcome: Percentage of Participants With Best Overall Response
Description: Best overall response according to IWCLL guidelines was defined as the percentage of patients with CR, CRi, PR or nodular Partial Response (nPR). CR required all of the following: Peripheral blood lymphocytes below 4 x 10^9/L, Absence of significant lymphadenopathy, No hepatomegaly, No splenomegaly, Absence of disease, Blood counts above the following values (Neutrophils >1.5 x 10^9/L, Platelets >100 x 10^9/L, Hemoglobin >11g/dL) and Bone marrow at least normocellular for age. CRi was CR with incomplete bone marrow recovery. PR required the following for at least 2 months from end of treatment: ≥50% decrease in peripheral blood lymphocyte count from the pre-treatment value AND Either a ≥ 50% reduction in lymphadenopathy OR ≥50% reduction of liver enlargement OR ≥50% reduction of spleen enlargement PLUS at least one of the following: Neutrophils >1.5 x 10^9/ or ≥50% increase, Platelets >100 x 10^9/L or ≥50% increase, Hemoglobin 11 g/dL or ≥50% increase.
Time Frame: Randomization to clinical cutoff (median observation 59.4 months)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab + Chlorambucil (RClb) | Obinutuzumab + Chlorambucil (GClb)
Number analyzed (Participants) | 330 | 333
percentage of participants
  Complete Response (CR) | 7.0 [4.5 to 10.3] | 23.7 [19.3 to 28.7]
  Complete Response incomplete (CRi) | 1.2 [0.3 to 3.1] | 1.8 [0.7 to 3.9]
  Partial Response (PR) | 55.5 [49.9 to 60.9] | 50.8 [45.2 to 56.2]
  Nodular Partial Response (nPR) | 2.7 [1.3 to 5.1] | 3.0 [1.4 to 5.5]
  Stable Disease | 14.5 [10.9 to 18.8] | 3.9 [2.1 to 6.6]
  Progressive Disease | 11.5 [8.3 to 15.5] | 4.5 [2.5 to 7.3]
  No Response Assessment | 7.6 [NA to NA] — 95% CI not estimated for No Response Assessment category. | 12.3 [NA to NA] — 95% CI not estimated for No Response Assessment category.
Statistical Analysis 1: Comparison: Rituximab + Chlorambucil (RClb) vs Obinutuzumab + Chlorambucil (GClb); Includes participants with best overall response: CR, CRi, PR or nPR; Test type: Superiority or Other; p = 0.0002, Chi-squared; Difference in Response Rates = 12.92, 95% CI 2-sided [6.1 to 19.8]

7. Secondary Outcome: Event Free Survival
Description: Event-free survival (EFS) was defined as the time between date of randomization and the date of disease progression/relapse, death, or start of a new anti-leukemic therapy. Progressive disease as per IWCLL criteria required at least one of the following: ≥50% increase in the absolute number of lymphocytes, appearance of new palpable lymph nodes (>15 mm in longest diameter) or any new extra nodal lesion, ≥50% increase in the longest diameter of any previous site of clinically significant lymphadenopathy, ≥50% increase in the enlargement of the liver and/or spleen, Transformation to a more aggressive histology or After treatment, the progression of any cytopenia (a decrease of hemoglobin levels >20 g/L or <10 g/dL or a decrease of platelet counts >50% or <100 x 10^9/L or by a decrease of neutrophil counts >50% or <1.0 x 10^9/L).
Time Frame: Randomization to clinical cutoff (median observation 59.4 months)
Population: ITT population included all randomized participants. Participants were censored at the date of last tumor assessment. In cases where no tumor assessment is available, participants were censored at the date of randomization plus one day.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab + Chlorambucil (RClb) | Obinutuzumab + Chlorambucil (GClb)
Number analyzed (Participants) | 330 | 333
months | 15 [14.2 to 17.1] | 26.5 [24.8 to 30.1]
Statistical Analysis 1: Comparison: Rituximab + Chlorambucil (RClb) vs Obinutuzumab + Chlorambucil (GClb); Test type: Superiority or Other; p < 0.0001, Log Rank, Stratified; Stratified by Binet stage at Baseline; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.43 to 0.61]

8. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) was defined as the time between the date of randomization and the date of death due to any cause.
Time Frame: Randomization to clinical cutoff (median observation 59.4 months)
Population: ITT population included all randomized participants. Participants who were not reported as having died at the time of the analysis were censored at the date when they were last known to be alive.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab + Chlorambucil (RClb) | Obinutuzumab + Chlorambucil (GClb)
Number analyzed (Participants) | 330 | 333
months | 73.1 [60.8 to NA] — The upper limit of 95% CI could not be estimated due to a low number of deaths. | NA [74.6 to NA] — The median overall survival and the upper limit of 95% CI could not be estimated due to a low number of deaths.
Statistical Analysis 1: Comparison: Rituximab + Chlorambucil (RClb) vs Obinutuzumab + Chlorambucil (GClb); Test type: Superiority or Other; p = 0.0245, Log Rank, Stratified; Stratified by Binet stage at Baseline; Hazard Ratio (stratified) = 0.76, 95% CI 2-sided [0.60 to 0.97]

9. Secondary Outcome: Duration of Response
Description: Duration of Response was defined as the date the response [either Complete Response (CR) or Partial Response (PR)] was first recorded until the date of Disease Progression or death due to any cause. Response was assessed according IWCLL guidelines.
Time Frame: Randomization to clinical cutoff (median observation 59.4 months)
Population: Participants from the ITT population, all randomized participants, with response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab + Chlorambucil (RClb) | Obinutuzumab + Chlorambucil (GClb)
Number analyzed (Participants) | 220 | 271
months | 11.8 [9.5 to 12.6] | 23.8 [19.1 to 30.1]
Statistical Analysis 1: Comparison: Rituximab + Chlorambucil (RClb) vs Obinutuzumab + Chlorambucil (GClb); Test type: Superiority or Other; p < 0.0001, Log Rank, Stratified; Stratified by Binet stage at Baseline; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.41 to 0.61]

10. Secondary Outcome: Percentage of Participants With Molecular Remission at the End of Treatment
Description: Molecular remission was defined as a minimal residual disease (MRD)-negative result at the end of treatment (assessment that occurred between 56 days and 6 months of last treatment). Molecular remission was assessed for all patients using a blood sample. Additionally, a bone marrow sample was obtained from patients whom the investigator assumed to have a complete response, consistent with the IWCLL guidelines. A combined analysis of blood and bone marrow results was conducted. A patient was considered MRD negative if result was less than 1 chronic lymphocytic leukemia (CLL) cell in 10000 leukocytes (MRD value < 0.0001) based on the method of allele specific polymerase chain reaction (ASO-PCR).
Time Frame: Randomization to clinical cutoff (median observation 59.4 months)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab + Chlorambucil (RClb) | Obinutuzumab + Chlorambucil (GClb)
Number analyzed (Participants) | 246 | 237
percentage of participants | 2 [0.9 to 5.2] | 24 [18.8 to 30.0]

11. Secondary Outcome: Time to Re-Treatment/New Anti-leukemic Therapy
Description: Time to re-treatment/new anti-leukemic therapy was defined as time between the date of randomization and the date of first intake of re-treatment or new anti-leukemic therapy.
Time Frame: Randomization to clinical cutoff (median observation 59.4 months)
Population: ITT population included all randomized participants. Participants who were reported as not having started re-treatment or new anti-leukemic therapy were censored at the last visit date they were assessed with regard to start of new treatment or the date of death.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab + Chlorambucil (RClb) | Obinutuzumab + Chlorambucil (GClb)
Number analyzed (Participants) | 330 | 333
months | 34.9 [29.1 to 41.6] | 56.4 [48.3 to NA] — Upper limit of 95% CI was not reached.
Statistical Analysis 1: Comparison: Rituximab + Chlorambucil (RClb) vs Obinutuzumab + Chlorambucil (GClb); Test type: Superiority or Other; p < 0.0001, Log Rank, Stratified; Stratified by Binet stage at Baseline; Hazard Ratio (stratified) = 0.58, 95% CI 2-sided [0.46 to 0.73]

12. Secondary Outcome: European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 Questionnaire
Description: The EORTC Quality of Life Questionnaire (QLQ-C30) was used to assess patient-reported outcomes (PRO) and symptom burden. The QLQ-C30 contains 30 items including the functional scales of physical functioning (5 items), role functioning (2 items), emotional functioning (4 items), cognitive functioning (2 items), social functioning (2 items) and symptom scales including fatigue (3 items), nausea and vomiting (2 items), and pain (4 items) and six single item scales on dyspnea, sleep disturbance, appetite loss, constipation, diarrhea and financial impact. Final scores are transformed such that they range from 0 - 100, whereby higher scores indicate greater functioning, greater quality of life, or a greater degree of symptoms, with changes of 5 - 10 points considered to be of minimally important difference to participants. A positive change from Baseline indicated improvement.
Time Frame: Baseline and Cycle 4 Day 1 (Cy4D1)
Population: ITT population. Here, n signifies the number of participants who were evaluated for specified category.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Rituximab + Chlorambucil (RClb) | Obinutuzumab + Chlorambucil (GClb)
Number analyzed (Participants) | 330 | 333
unit on a scale
  Appetite Loss Scale: Baseline (n=314, 312) | 15.4 (26.02) | 19 (29.37)
  Appetite Loss Scale: Cy4D1 (n=277, 258) | 12 (23.22) | 10.9 (21.47)
  Cognitive Functioning Scale: Baseline(n=312, 315) | 83.0 (20.02) | 80.4 (22.52)
  Cognitive Functioning Scale: Cy4D1 (n=277, 259) | 83.6 (17.26) | 83.9 (20.25)
  Constipation Scale: Baseline (n=311, 312) | 15.2 (24.62) | 14.9 (23.54)
  Constipation Scale: Cy4D1 (n=276,257) | 14.3 (23.05) | 15.3 (25.16)
  Diarrhoea Scale: Baseline (n=311,313) | 8.4 (18.78) | 9.5 (19.58)
  Diarrhoea Scale: Cy4D1 (n=276,257) | 8.8 (19.66) | 9.2 (20.32)
  Dyspnoea Scale: Baseline (n=312,312) | 27.5 (28.62) | 27.8 (29.97)
  Dyspnoea: Cy4D1 (n=277,257) | 20.8 (26.69) | 16.5 (23.75)
  Emotional Functioning Scale: Baseline (n=312,314) | 77.1 (21.32) | 73.9 (23.14)
  Emotional Functioning Scale: Cy4D1 (n=277,259) | 82.7 (18.29) | 82.5 (19.18)
  Fatigue Scale: Baseline (n=313,312) | 36.9 (25.86) | 38.5 (26.05)
  Fatigue Scale: Cy4D1 (n=278,258) | 30.4 (22.32) | 29.8 (21.43)
  Financial Difficulties Scale: Baseline (n=309,312) | 10.5 (21.53) | 10.5 (22.14)
  Financial Difficulties Scale: Cy4D1(n=273,258) | 9.6 (20.02) | 8.4 (19.35)
  Nausea, Vomiting Scale: Baseline (n=313,315) | 4.5 (12.66) | 5.3 (12.9)
  Nausea, Vomiting Scale: Cy4D1 (n=278,258) | 4.1 (10.18) | 5.2 (10.96)
  Pain scale: Baseline (n=313,316) | 22.5 (27.59) | 22.9 (27.73)
  Pain scale: Cy4D1 (n=278,259) | 15.6 (22.48) | 18.1 (24.60)
  Physical Functioning Scale: Baseline (n=313,316) | 75.8 (19.34) | 73.3 (20.77)
  Physical Functioning Scale: Cy4D1 (n=278,258) | 77.8 (18.5) | 78.5 (18.90)
  Global Health Status Scale: Baseline (n=310,313) | 58.1 (22.74) | 58.0 (23.81)
  Global Health Status Scale: Cy4D1 (n=275,256) | 65.8 (20.22) | 66.7 (20.27)
  Role Functioning Scale: Baseline (n=313,315) | 76.4 (28.68) | 74.3 (27.62)
  Role Functioning Scale: Cy4D1 (n=277,258) | 79.9 (25.4) | 78.7 (24.56)
  Social Functioning Scale: Baseline (n=312,314) | 82.9 (23.81) | 83.7 (24.96)
  Social Functioning Scale: Cy4D1(n=276,259) | 85.4 (21) | 86.6 (20.71)
  Insomnia: Baseline (n=312,316) | 25.6 (30.91) | 29.9 (31.18)
  Insomnia: Cy4D1(n=276,258) | 20.9 (26.71) | 21.6 (27.97)

13. Secondary Outcome: European Organization for Research and Treatment of Cancer (EORTC) QLQ-CLL16 Questionnaire
Description: EORTC Quality of Life Questionnaire (QLQ-CLL16) module was used to assess patient-reported outcomes and symptom burden. The QLQ-CLL16 module includes three multi-item scales assessing fatigue (2 items), treatment side effects and disease symptoms (8 items), infection (4 items) and two single item scales on social activities and future health worries. Final scores are transformed such that they range from 0 - 100, whereby higher scores indicate greater functioning, greater quality of life, or a greater degree of symptoms, with changes of 5 - 10 points considered to be of minimally important difference to participants. A positive change from Baseline indicated improvement.
Time Frame: Baseline and Cycle 4 Day 1 (Cy4D1)
Population: ITT population. Here, n signifies the number of participants who were evaluated for specified category.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Rituximab + Chlorambucil (RClb) | Obinutuzumab + Chlorambucil (GClb)
Number analyzed (Participants) | 330 | 333
unit on a scale
  Disease Effects Scale: Baseline (n=276,284) | 22.8 (17.94) | 22.7 (18.49)
  Disease Effects Scale: Cy4D1 (n=243, 233) | 15.4 (15) | 14.7 (15.34)
  Fatigue Scale: Baseline (n=276, 284) | 27.7 (23.48) | 31.1 (25.32)
  Fatigue Scale: Cy4D1 (n=243, 233) | 21 (20.52) | 20.6 (20.82)
  Future Health: Baseline (n=275, 280) | 47.5 (32.17) | 49.8 (32.79)
  Future Health: Cy4D1 (n=240, 231) | 33.9 (29.72) | 30.3 (31.17)
  Infection Scale: Baseline (n=275, 284) | 11.8 (15.83) | 12.7 (16.67)
  Infection Scale: Cy4D1 (n=243, 233) | 9.4 (13.94) | 9 (12.2)
  Social Problems: Baseline (n=271, 281) | 25.2 (32.45) | 23.6 (31.12)
  Social Problems: Cy4D1 (n=242, 232) | 19.3 (26.03) | 19.5 (27.94)
  Treatment Side Effects Scale: Baseline(n=276, 284) | 17.9 (15.69) | 19.9 (17.59)
  Treatment Side Effect Scale: Cy4D1(n=243, 233) | 14.2 (13.57) | 14.6 (14.89)

ADVERSE EVENTS:
Time Frame: 5.5 years
Description: Safety Population included all randomized participants who received at least one dose of study drug. 4 patients randomized to RClb and 2 patients randomized to GClb did not receive study drug. In addition, 5 participants in the RClb arm received at least 1 dose of obinutuzumab and are included in the GClb arm for safety analyses.
Arm/Group | Rituximab + Chlorambucil (RClb) | Obinutuzumab + Chlorambucil (GClb)
Serious Adverse Events (participants affected / at risk) | 124/321 | 150/336
Other Adverse Events (participants affected / at risk) | 279/321 | 299/336
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Chlorambucil (RClb) (N=321) | Obinutuzumab + Chlorambucil (GClb) (N=336)
Pneumonia (Infections and infestations) | 19 | 14
Respiratory tract infection (Infections and infestations) | 2 | 3
Bronchitis (Infections and infestations) | 3 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 3
Neutropenic sepsis (Infections and infestations) | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 1
Urinary tract infection (Infections and infestations) | 1 | 3
Cellulitis (Infections and infestations) | 3 | 0
Infection (Infections and infestations) | 2 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Endocarditis (Infections and infestations) | 1 | 1
Erysipelas (Infections and infestations) | 0 | 2
Escherichia infection (Infections and infestations) | 1 | 1
Hepatitis B (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 0 | 2
Streptococcal sepsis (Infections and infestations) | 1 | 1
Varicella (Infections and infestations) | 2 | 0
Wound infection (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 1 | 0
Dacryocystitis (Infections and infestations) | 0 | 1
Device related sepsis (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis clostridial (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0
Infectious colitis (Infections and infestations) | 0 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 1
Intervertebral discitis (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 1
Septic arthritis staphylococcal (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1
Superinfection bacterial (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 6
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 8
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 4
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 34
Fall (Injury, poisoning and procedural complications) | 1 | 3
Femur fracture (Injury, poisoning and procedural complications) | 3 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 2
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
Shunt thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 6
Neutropenia (Blood and lymphatic system disorders) | 2 | 4
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 4
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 2
Pancytopenia (Blood and lymphatic system disorders) | 2 | 1
Cytopenia (Blood and lymphatic system disorders) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 4
Myocardial infarction (Cardiac disorders) | 0 | 4
Atrial fibrillation (Cardiac disorders) | 1 | 2
Cardiac arrest (Cardiac disorders) | 3 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Nodal rhythm (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Death (General disorders) | 3 | 0
Pyrexia (General disorders) | 2 | 2
Chest pain (General disorders) | 2 | 1
General physical health deterioration (General disorders) | 3 | 1
Asthenia (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 2 | 0
Adhesion (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Impaired healing (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Colitis (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 3
Central nervous system haemorrhage (Nervous system disorders) | 0 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Capillary leak syndrome (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Diabetic macroangiopathy (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Malignant hypertension (Vascular disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Nephritic syndrome (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 1 | 0
Mania (Psychiatric disorders) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Hereditary non-polyposis colorectal cancer syndrome (Congenital, familial and genetic disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Testicular hypertrophy (Reproductive system and breast disorders) | 0 | 1
Hepatitis B Reactivation (Infections and infestations) | 1 | 0
Basosquamous Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant Melanoma in Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Polycythaemia Vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Chlorambucil (RClb) (N=321) | Obinutuzumab + Chlorambucil (GClb) (N=336)
Neutropenia (Blood and lymphatic system disorders) | 104 | 128
Anaemia (Blood and lymphatic system disorders) | 34 | 33
Thrombocytopenia (Blood and lymphatic system disorders) | 20 | 46
Leukopenia (Blood and lymphatic system disorders) | 7 | 21
Infusion related reaction (Injury, poisoning and procedural complications) | 118 | 197
Nausea (Gastrointestinal disorders) | 42 | 40
Diarrhoea (Gastrointestinal disorders) | 24 | 31
Constipation (Gastrointestinal disorders) | 16 | 27
Vomiting (Gastrointestinal disorders) | 22 | 19
Fatigue (General disorders) | 30 | 26
Pyrexia (General disorders) | 22 | 28
Asthenia (General disorders) | 25 | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 24
Headache (Nervous system disorders) | 18 | 23
Rash (Skin and subcutaneous tissue disorders) | 19 | 8
Urinary Tract Infection (Infections and infestations) | 6 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.